CLINICAL TRIAL: NCT06368284
Title: Observational Study of Perineal Trauma After Jet Ski Accidents and Long-term Functional Outcomes Results
Brief Title: Perineal Trauma After Jet Ski Accidents and Long-term Functional Outcomes Results
Acronym: TP-JET
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-MTP_2022_09_202201170
Record Dates: First submitted 2024-04-05; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Perineum; Tear, Traumatic; Anal Tear; Anal Incontinence
Keywords: Ano-perineal trauma; Ano-perineal injury; Personal watercraft; Jet-Ski; functional outcomes; peripheral neurogenic bladder; fecal incontinence
MeSH Terms: conditions — Lacerations; Encopresis; Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Patients who experienced an ano-perineal trauma following a PWC/Jet-Ski accident — Patients who experienced an ano-perineal trauma following a PWC/Jet-Ski accident between January 2017 and December 2023, managed and followed up in France

SUMMARY:
French multicentric retrospective cohort study including patients who underwent an ano-perineal trauma following a personal watercraft/jet-ski accident and that were treated in France from January 2017 to December 2023.

Aims of the study were to describe the initial management of the patients and to evaluate the digestive, urological and sexual functional outcomes as well as the quality of life, using validated questionnaires commonly employed in clinical practice.

DETAILED DESCRIPTION:
Ano-perineal injuries and their mechanisms resulting from personal watercraft (PWC)/Jet-Ski accidents are poorly understood and may lead to long-term functional repercussions, previously unmentioned in studies. These accidents are in France but, mostly, concerned young women, back-seated on the PWC without any specific protection.

Therefore, the research team conducted a French multicentric cohort study that retrospectively included patients who experienced ano-perineal trauma following a personal watercraft/Jet-Ski accident and were treated in France.

Data on pre-hospital management, pre-operative work-up, surgical management (including surgical techniques), short-term and long-term complications (routinely used functional scores) were collected through the analysis of personal medical records.

Several patients had sphincteric, rectal, vaginal, or combined injuries, sometimes requiring the establishment of a stoma. the investigators subsequently evaluated the rate of fecal incontinence (evaluated by anorectal manometry or Wexner score), urological (USP score), and sexual outcomes (FSFI). Quality of life was also assessed using the SF12 score.

ELIGIBILITY:
Inclusion Criteria:

* ano-perineal trauma following a PWC/Jet-Ski accident between January 2017 and December 2023
* managed and followed in France

Exclusion Criteria:

* <18 years old

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who experienced an ano-perineal trauma following a PWC/Jet-Ski accident between January 2017 and December 2023, managed and followed up in France
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of fecal incontinence | Consultation at 12 months of trauma on average
  Defined by the fecal incontinence Wexner Score >10 (Score from 0 to 20, the higher the score, the greater the incontinence.) or by ano-rectal manometry.

SECONDARY OUTCOMES:
Rate of permanent stoma | Consultation at 12 months of trauma on average
  No long-term plan for restoration of digestive continuity
Rate of acontractile bladder | Consultation at 12 months of trauma on average
  Self-catheterization
Rate of sexual dysfunction | Consultation at 12 months of trauma on average
  defined as Female Sexual Function Index (FSFI) score <26,55 (Score from 2 to 36, the lower the score, the greater the dysfunction.)
Rate of impact on quality of life | Consultation at 12 months of trauma on average
  rated by 12-Item Short Form Survey (SF-12) (the higher the score, the greater the quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas BARDOL, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Chu Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No